CLINICAL TRIAL: NCT00478816
Title: A Phase II, Single Center, Exploratory Study to Evaluate Safety and Immunogenicity of Two Doses of H5N1 Influenza Vaccine in Adults Unprimed and Primed With MF59-adjuvanted or Non-adjuvanted H5N3 Influenza Vaccines
Brief Title: Safety and Immunogenicity of Two Doses of H5N1 Influenza Vaccine in Adults Unprimed and Primed With Adjuvanted or Non-adjuvanted Influenza Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V87P3
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-02

CONDITIONS: Prophylaxis of Avian Influenza Vaccine
Keywords: Bird flu; influenza vaccine; prepandemic vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Primed subject with pandemic Vaccine
  Interventions: Biological: Fluad H5N1 Pandemic Influenza Vaccine
- Group 2 (Active Comparator): Non Primed subject with pandemic Vaccine
  Interventions: Biological: Fluad H5N1 Pandemic Influenza Vaccine

INTERVENTIONS:
Biological: Fluad H5N1 Pandemic Influenza Vaccine — Two 0.5 mL doses of MF59-adjuvanted A/Vietnam/1194/2004 (H5N1 Clade 1) hemagglutinin (HA) subvirion influenza vaccine, containing 7.5 μg of H5N1 antigen,administered 3 weeks apart, IM in the deltoid muscle, preferably of the non-dominant arm.
  Other Names: Vaccine

SUMMARY:
Valuate the immune response and reactogenicity of H5N1 vaccination in a primed population (H5N3 adjuvanted or non-adjuvanted vaccine) compared to immunologically naïve subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 65 years of age, mentally competent, who have signed an informed consent form after having received a detailed explanation of the study protocol;
2. In good health as determined by:

   1. medical history,
   2. physical examination,
   3. clinical judgment of the Investigator;
3. Subjects in the primed group previously received at least two doses of an H5N3 vaccine;
4. Able to understand and comply with all study procedures and to complete study diaries, can be contacted, and will be available for study visits.

Exclusion Criteria:

1. Receipt of another investigational agent within 4 weeks, or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another clinical study through the end of the study;
2. Subjects who experienced any acute disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) within the past 7 days;
3. Subjects who experienced fever (defined as axillary temperature ≥38.0°C) within 3 days prior to Visit 1;
4. Subjects who are pregnant or breastfeeding;
5. Females of childbearing potential who refuse to use an acceptable method of birth control for the duration of the study. Adequate contraception is defined as hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom with spermicide or diaphragm with spermicide), intrauterine device (e.g., IUD), or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry;
6. Subjects with any serious disease, such as:

   1. cancer,
   2. autoimmune disease (including rheumatoid arthritis),
   3. diabetes mellitus,
   4. chronic pulmonary disease,
   5. acute or progressive hepatic disease,
   6. acute or progressive renal disease;
7. Subjects for whom a surgery is planned during the study period;
8. Subjects with bleeding diathesis;
9. Subjects with hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the study vaccine;
10. Subjects with a history of any neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
11. Subjects with known or suspected impairment/alteration of immune function, for example, resulting from:

    1. receipt of immunosuppressive therapy (any corticosteroid therapy or cancer chemotherapy),
    2. receipt of immunostimulants,
    3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Visit 1 or planned during the full length of the study,
    4. high risk for developing an immunocompromising disease;
12. Receipt of another vaccine within 3 weeks prior to Visit 1 or planned vaccination within 3 weeks following the last study vaccination;
13. Subjects with a history of (or current) drug or alcohol abuse that in the investigator's opinion would interfere with safety of the subject or the evaluation of study objectives;
14. Subjects with any condition, which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Cell-mediated immunity, magnitude, breath and kinetics of antibody response to 2 doses of MF59-adjuvanted H5N1 influenza vaccine, in subjects primed by previous vaccination with either MF59-adjuvanted or non-adjuvanted H5N3 influenza vaccine. | Days 1, 8, 15, 22, 43 and 202

SECONDARY OUTCOMES:
Safety Objectives: safety and reactogenicity of the vaccine | Days 1, 8, 15, 22, 43 and 202

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines Information Service +41 61 324 1111, Study Chair — Novartis
Locations (1):
- Infectious Diseases Unit, Leicester, United Kingdom

REFERENCES:
- [Result] Galli G, Hancock K, Hoschler K, DeVos J, Praus M, Bardelli M, Malzone C, Castellino F, Gentile C, McNally T, Del Giudice G, Banzhoff A, Brauer V, Montomoli E, Zambon M, Katz J, Nicholson K, Stephenson I. Fast rise of broadly cross-reactive antibodies after boosting long-lived human memory B cells primed by an MF59 adjuvanted prepandemic vaccine. Proc Natl Acad Sci U S A. 2009 May 12;106(19):7962-7. doi: 10.1073/pnas.0903181106. Epub 2009 Apr 27. PMID 19416838